CLINICAL TRIAL: NCT02009124
Title: Open Label Study of Autologous Bone Marrow Mononuclear Cells in Spinal Cord Injury
Brief Title: Stem Cell Therapy in Spinal Cord Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-03
Record Dates: First submitted 2013-12-02; First posted 2013-12-11 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; stem cell therapy; bone marrow; mononuclear cells; autologous
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem cell (Experimental): autologous bone marrow mononuclear cell transplantation
  Interventions: Biological: Autologous bone marrow mononuclear cell transplantation
- Control (No Intervention): Stem cell therapy is not done for this group of spinal cord injury patients

INTERVENTIONS:
Biological: Autologous bone marrow mononuclear cell transplantation — Bone marrow is aspirated by a standard procedure. Mononuclear cells are separated by density gradient method and then injected intrathecally by a standard lumbar puncture procedure
  Arms: Stem cell

SUMMARY:
The purpose of this study is to study the effect of stem cell therapy on common symptoms in patients with spinal cord injury.

DETAILED DESCRIPTION:
Autologous bone marrow mononuclear cells are administered intrathecally by a standard procedure followed by vigorous rehabilitation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of any type of spinal cord injury
* age above 12 months.

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* space occupying lesion in brain
* other acute medical conditions such as respiratory infection and pyrexia.

Ages: 12 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in clinical symptoms of spinal cord injury after 6 months | 6 months

SECONDARY OUTCOMES:
Functional independence measure (FIM) | 6 months
  It is a standard objective scale used for functional evaluation of the spinal cord injury patients. Its reliability and validity has been well established. It will be marked by a certified occupational therapy expert before the intervention and 6 months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alok K Sharma, MS,MCh, Principal Investigator — Neurogen Brain and Spine Institute
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Sharma A, Gokulchandran N, Sane H, Badhe P, Kulkarni P, Lohia M, Nagrajan A, Thomas N. Detailed analysis of the clinical effects of cell therapy for thoracolumbar spinal cord injury: an original study. Journal of Neurorestoratology. 2013;1:13-22
- [Background] Sharma A, Sane H, Gokulchandran N, Kulkarni P, Thomas N, et al. (2013) Role of Autologous Bone Marrow Mononuclear Cells in Chronic Cervical Spinal Cord Injury-A Longterm Follow Up Study. J Neurol Disord 1: 138.
- [Background] Kumar AA, Kumar SR, Narayanan R, Arul K, Baskaran M. Autologous bone marrow derived mononuclear cell therapy for spinal cord injury: A phase I/II clinical safety and primary efficacy data. Exp Clin Transplant. 2009 Dec;7(4):241-8. PMID 20353375
- [Background] Yoshihara T, Ohta M, Itokazu Y, Matsumoto N, Dezawa M, Suzuki Y, Taguchi A, Watanabe Y, Adachi Y, Ikehara S, Sugimoto H, Ide C. Neuroprotective effect of bone marrow-derived mononuclear cells promoting functional recovery from spinal cord injury. J Neurotrauma. 2007 Jun;24(6):1026-36. doi: 10.1089/neu.2007.132R. PMID 17600518
- [Background] Sharma A, Gokulchandran N, Chopra G, Kulkarni P, Lohia M, Badhe P, Jacob VC. Administration of autologous bone marrow-derived mononuclear cells in children with incurable neurological disorders and injury is safe and improves their quality of life. Cell Transplant. 2012;21 Suppl 1:S79-90. doi: 10.3727/096368912X633798. PMID 22507683